CLINICAL TRIAL: NCT01883648
Title: A Randomized, Double-Blind, Placebo-Controlled, 6 Month Cross-Over Study to Evaluate the Efficacy of Coconut Oil (Fuel for Thought™) Treatment for Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Study to Evaluate Coconut Oil for Alzheimer's Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding limitations and enrollment was too low.
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Byrd AD-001
Record Dates: First submitted 2013-06-11; First posted 2013-06-21 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: Mild to Moderate Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coconut Oil Beverage (Experimental): The treatment will consist of a 1.25 oz serving size taken orally, two times daily by subjects. This treatment arm will last 3 months.
  Interventions: Drug: Coconut Oil Beverage
- Placebo Beverage (Placebo Comparator): The treatment will consist of a 1.25 oz serving size taken orally, two times daily by subjects.This will similar in look and taste but not have the same ingredients of the actual coconut oil beverage. This treatment arm will last 3 months.
  Interventions: Other: Placebo Beverage

INTERVENTIONS:
Drug: Coconut Oil Beverage — There are 2 treatment arms: Fuel for Thought™ and placebo, with a treatment allocation of 1:1. After 3 months of treatment in one group, subjects will have a 3-5 day wash-out period before receiving the alternate (opposite) treatment for 3 months.
  Other Names: Fuel for Thought (TM)
  Arms: Coconut Oil Beverage
Other: Placebo Beverage — There are 2 treatment arms: Fuel for Thought™ and placebo, with a treatment allocation of 1:1. After 3 months of treatment in one group, subjects will have a 3-5 day wash-out period before receiving the alternate (opposite) treatment for 3 months.
  Arms: Placebo Beverage

SUMMARY:
This is a randomized, cross over study to determine the efficacy of coconut oil in subjects with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, cross over study to determine the efficacy of coconut oil (a proprietary blend of coconut and medium chain triglyceride oils, administered orally three times daily) to subjects with Alzheimer's disease who have been screened for ApoE 4 allele. The study medication formula is Cognate Nutritionals Fuel for Thought™.

Approximately 65 subjects will be treated with a coconut oil beverage (Fuel for Thought™) or placebo for three months, and then given a 3-5 day interim wash out period. After this, subjects will resume with three months treatment in opposite treatment arm. Total treatment period is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 55 to 90 years with a diagnosis of mild to moderate Alzheimer's disease
* Informed consent signed and dated by subject (or legally authorized representative).
* Subjects must have a study partner must also consent to participate in the study, who they spend at least 10 hours/week with during the study. The study partner must attend applicable clinic visits and provide information about the subject.
* Subject must have a screening Mini-Mental State Examination score of 16-26.
* Subjects must have a Rosen Modified Hachinski Ischemic score of ≤4.
* Subject must undergo ApoE genetic laboratory testing at the baseline visit.
* Subject must be willing and able to take study medication (or placebo) for the duration of the study.
* Subject must be stable on all memory enhancing medications including cholinesterase inhibitors (including donepezil, rivastigmine, and galantamine) and NMDA antagonist (memantine) for at least 3 months prior to screening and agree not to change these medications during the course of their participation, unless medically necessary.
* Subject must be stable on all memory enhancing nonprescription supplements (including gingko biloba, huperzine, resveratrol, or docosahexaenoic acid) for at least 3 months prior to screening and agree not to change these medications during the course of their participation.
* As judged by Investigator, the subject and study partner will be compliant and have a high probability of completing the study, including all scheduled evaluations and required tests.
* Be fluent in English.

Exclusion Criteria:

* Has significant neurological or medical disease, other than AD, that may affect cognition, for example, history or evidence of hydrocephalus, or uncontrolled hypo- or hyperthyroidism.
* Current, clinically significant major psychiatric disorder (eg, major depressive disorder) according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSMIV), or symptoms (eg, hallucinations) that could affect the subject's ability to complete the study.
* Geriatric depression scale score of more than 6 or has suicidal ideation.
* Current clinically significant chronic illness that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study, including uncontrolled diabetes. Subjects with a history of diabetic ketoacidosis will also be excluded. Other cases of diabetes will be decided at the discretion of the study physicians. Subjects with diabetes controlled with exercise and diet may be screened and admission to study will depend on their screening safety laboratory assessments.
* History of clinically evident stroke or history of clinically significant carotid or vertebrobasilar stenosis or plaque and other risk factors for thromboembolic stroke (e.g atrial fibrillation, clinically significant low ventricular output, atrial septal defect).
* History of seizures.
* Clinically significant infection within the last 30 days (eg, chronic persistent or acute infection [eg, upper respiratory infection, urinary tract infection]),prior to screening.
* Myocardial infarction within the last 2 years.
* Abnormal screening visit electrocardiogram (ECG), in the opinion of the investigator.
* Uncontrolled hypertension within the last 6 months prior to screening.
* History of cancer within the last 3 years, with the exception of nonmetastatic basal cell carcinoma and squamous cell carcinoma of the skin. (Note: cancer must be in remission with no signs of progression.)
* Use of experimental or other investigational medications/devices for treatment within 90 days prior to screening.
* Laboratory findings of fasting total cholesterol greater than or equal to 240 mg/dL
* Laboratory findings of fasting triglycerides greater than or equal to 200 mg/dL
* Laboratory findings of fasting glucose greater than or equal to 126 mg/dL
* Other clinically significant abnormality on physical, neurological, laboratory, vital signs, or ECG examination (eg, changes consistent with recent infarction, ischemia, clinically significant arrhythmias and clinically significant conduction defects) that could be detrimental to the subject or compromise the study.
* Does not have adequate venous access that would allow blood draws.
* Subject or study partner is related to study personnel.
* Subjects who have taken coconut oil as a supplement within the last 30 days.
* Subjects who have taken Axona™ within the last 30 days.
* Women who are pregnant. (Women who are of child bearing potential must take precautions to not become pregnant during the study.)

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in cognitive testing (ADAS-cog, MMSE, Category/Letter Fluency) | Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in cognitive testing (ADAS-cog, MMSE, Category/Letter Fluency)

SECONDARY OUTCOMES:
Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in Trails A & B cognitive testing | Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in Trails A & B cognitive testing
Change from baseline to Month 3 of each treatment phase (a 3 month period of time) on Geriatric Depression Scale | Change from baseline to Month 3 of each treatment phase (a 3 month period of time) on Geriatric Depression Scale
Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in behaviors measured by Neuropsychiatric Inventory | Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in behaviors measured by Neuropsychiatric Inventory
Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in functional ability measured by Activities of Daily Living (ADCS-ADLs) | Change from baseline to Month 3 of each treatment phase (a 3 month period of time) in functional ability measured by Activities of Daily Living (ADCS-ADLs)
Measure changes in Ketone & C-Reactive Protein assays from research blood samples throughout study during the 2 treatment periods from Baseline to Month 6 (change during a total 6 month period of time). | Measure changes in Ketone & C-Reactive Protein assays from research blood samples throughout study during the 2 treatment periods from Baseline to Month 6 (change during a total 6 month period of time).
Adverse events related to coconut oil usage during 6 months of treatment periods (change during a total 6 month period of time). | Adverse events related to coconut oil usage during 6 months of treatment periods (change during a total 6 month period of time).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda G Smith, MD, Principal Investigator — USF Health Byrd Alzheimer's Institute
Locations (1):
- USF Health Byrd Alzheimer's Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No